CLINICAL TRIAL: NCT05117710
Title: Does the IMPase Inhibitor, Ebselen, Affect Emotional Processing and Brain Myo-inositol in Treatment-resistant Depression?
Brief Title: IMPase in Treatment-resistant Depression
Acronym: OxIMP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 276211; 20/SC/0151 (Other: South Central Oxford B REC)
Record Dates: First submitted 2021-09-13; First posted 2021-11-11 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Treatment Resistant Depression; Ebselen
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — ebselen

STUDY DESIGN:
Intervention Model Description: Parallel-arm, double-blind, randomised, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ebselen (Active Comparator): The intervention will be 7-10 days administration of ebselen 600 mg twice daily taken orally. Ebselen has been manufactured to Good Manufacturing Practice (GMP) standards and will be provided by Sound Pharmaceuticals Inc. in 200 mg capsules.
  Interventions: Drug: Ebselen
- Placebo (Placebo Comparator): The intervention will be 7-10 days administration of placebo 600 mg twice daily taken orally.Identical placebo capsules have been manufactured and formulated in the same facilities as the active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ebselen — Ebselen is an organoselenium compound, developed originally as an antioxidant for use in neuroprotection, post-stroke. Ebselen is a bioavailable and brain penetrant inhibitor of inositol monophosphatase (IMPase) (Ki ≈ 1 μM).
  Other Names: SPI-1005; PZ-51; Ebselene; Ebselenum; Ebseleno; Harmokisane
  Arms: Ebselen
Drug: Placebo — Matched placebo capsules
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
This experimental medicine study will examine the effects of a brief period (seven days) of 'add on' ebselen (SPI-105) treatment in patients with resistant depression to see if ebselen produces changes in emotional responses consistent with a potential clinical antidepressant effect. The investigators will also seek to confirm ebselen's mode of action on IMPase by measuring changes in a brain chemical called inositol, using a magnetic imaging method. Half of the participants will receive ebselen and the other half placebo.

DETAILED DESCRIPTION:
Ebselen, a potential new drug for treatment resistent depression (TRD).

Clinical depression is an important public health problem, associated with an even greater burden of illness than other common diseases such as angina, arthritis, asthma, and diabetes. The burden of illness is particularly high for depressed patients in specialist psychiatric care who often fare poorly with current treatments and who typically experience substantial functional disability with a significantly increased risk of suicide. A limiting factor in improving outcome for such patients is the lack of acceptable pharmacological approaches for so-called 'TRD'. In a recent large randomised trial, even specialist mood disorder services with access to expert psychological and pharmacological treatment, struggled to improve therapeutic response rates compared to 'treatment as usual'. This indicates that improving the management of TRD requires more than improved access to specialist clinics - new, more effective and better tolerated therapies are needed.

The principal aim of the current study is to examine the utility of a potential new lithium-mimetic drug, ebselen, in patients with TRD. Lithium itself is known to be efficacious in the management of TRD as an 'add-on' treatment to ineffective antidepressant medication. However, its poor tolerability and safety and the need for regular blood tests has resulted in it having a low acceptability for both patients and clinicians.

Lithium has many pharmacological targets but inhibition of an enzyme called inositol monophosphatase (IMPase) is an important candidate for its therapeutic effects in mood disorders. However, this potential mechanism has not been tested previously in depressed patients. Ebselen is an organoselenium compound, developed originally as an antioxidant for use in neuroprotection, post-stroke. Although clinical trials indicated that ebselen was safe and well-tolerated, its therapeutic activity in stroke patients was limited and its commercial development was halted. Subsequent work in the University of Oxford's Department of Pharmacology found that ebselen is a bioavailable and brain penetrant inhibitor of inositol monophosphatase (IMPase) (Ki ≈ 1 μM) (8). This finding provides an opportunity to use ebselen as a means of testing the role of IMPase inhibition in the therapeutic effect of lithium in TRD.

Recently, experimental medicine models developed in the University of Oxford's Department of Psychiatry have shown promise in describing early surrogate markers of patient responsiveness to antidepressants. Traditionally, the translation of novel potential antidepressant compounds from animal studies to humans has involved placebo-controlled clinical trials that are expensive and take many years. The newer, more experimental medicine studies exploiting the use of surrogate markers for depression and antidepressant drug action have the potential to transform this field and refine development decisions while minimising time and cost and burden on patients.

The surrogate markers of antidepressant efficacy that the investigators have developed for this process are based on cognitive theories of depression and antidepressant action. Cognitive theories of depression outline the role of negative emotional biases in information processing in the aetiology and maintenance of the disorder. For example, compared to controls, depressed patients are more likely to perceive ambiguous facial expressions as negative and to retrieve negative self-relevant information in both explicit and indirect memory paradigms. These cognitive biases are believed to play a key role in the persistence of the depressed state because increased accessibility of negative perceptions and memories maintains and exaggerates the depressed mood leading to a self-perpetuating cycle.

Importantly, cognitive biases shift early in antidepressant treatment, and positive changes in emotional processing can be demonstrated in relatively small groups of patients. Subsequent studies showed that early positive shifts in emotional processing predict eventual therapeutic outcome to antidepressant medication.

The investigators have previously used these experimental medicine approaches to assess the effects of ebselen in healthy volunteers. The investigators found that, given at a dose of 600 mg, as well as 1200 mg twice daily, ebselen produced a greater recognition of some positive emotions, an effect the investigators have noted with numerous typical and atypical antidepressants and a strong predictor of clinical antidepressant activity. The investigators also utilised magnetic resonance spectroscopy (MRS), and demonstrated a reduction in brain inositol after treatment with ebselen. This provides evidence for IMPase target engagement of ebselen at the dose proposed for this study. Therefore, the investigators now have substantial data that indicates that ebselen is a valid means of testing IMPase inhibition as a potential antidepressant mechanism in a clinical population of TRD patients, using an experimental medicine approach.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study;
* Sufficiently fluent English to understand and complete the tasks;
* Registered with a General Practitioner (GP) and consents to GP being informed of participation in the study;
* Participants need to meet a number of concurrent clinical criteria:
* Current criteria for Major Depressive Disorder as determined by the Structured Clinical Interview for Diagnostic and Statistical Manual-5 (SCID-5);
* Inadequate response to at least one adequate course of antidepressant therapy given at a therapeutic dose for at least four weeks in the current episode of depression.
* Minimum score on the 17-item Hamilton Depression Rating Scale (HAM-D) of at least 14;
* Currently taking a licensed antidepressant at a therapeutic dose for at least four weeks
* Pre-menopausal women and male participants engaging in sex with a risk of pregnancy must agree to use a highly effective method of contraception from Screening Visit until 30 days after receiving the study medication treatment. Acceptable methods of contraception include:

  * Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal or transdermal;
  * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable or implantable;
  * Intrauterine device (IUD);
  * Intrauterine hormone-releasing system (IUS);
  * Bilateral tubal occlusion;
  * Vasectomy (or vasectomised partner);
  * Sexual abstinence. [Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), and spermicides only are not acceptable methods of contraception.]
* Male participants must not donate sperm.
* Participants taking non-prescription/prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety
* Willing to refrain from drinking alcohol for the duration of the study

Exclusion Criteria:

* History of /or current DSM-5 bipolar disorder, schizophrenia or emotionally unstable personality disorder;
* Participants who fulfil current criteria for other comorbid disorders may still be entered into the study, if, in the opinion of the Investigator, the psychiatric diagnosis will not compromise safety or affect data quality;
* Participants who have failed to respond to standard pharmacological augmentation treatments for depression (lithium and atypical antipsychotic drugs);
* Clinically significant risk of suicide;
* Participants undergoing or who have undergone electroconvulsive therapy for the treatment of the current episode of depression;
* History of significant alcohol/substance misuse or dependence over the past 6 months;
* History of, or current general medical conditions that in the opinion of the Investigator may interfere with the safety of the participant or the scientific integrity of the study;
* Current pregnancy (as determined by urine pregnancy test taken during the Screening Visit and the Research Visit One), breastfeeding, or planning a pregnancy during the course of the study;
* Participants with Body Mass Index (BMI - kg/m2) outside the 18-36 range at Screening Visit;
* Participants with severe claustrophobia;
* Participants who are contraindicated for MRI;
* Previous participation in a study using the same, or similar, emotional processing tasks in the last three months;
* Previous participation in a study involving the use of an interventional medication within the last three months;
* Participant with planned medical treatment within the study period that might interfere with the study procedures;
* Participant who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in positive and negative facial expression recognition task | Change between groups from baseline to day 7
  Difference in accuracy to recognise computer-based positive and negative facial expressions (anger, disgust, fear, happy, sad, surprise)
Change in misclassifications on emotional processing task | Change between groups from baseline to day 7
  Differences in misclassifications (number of responses to each facial expression category incorrectly classified as another facial expression category).
Change in reaction time on emotional processing task | Change between groups from baseline to day 7
  Differences in reaction time to recognise facial expressions

SECONDARY OUTCOMES:
Change in accuracy in the Emotional Categorisation Task | Change between groups from baseline to day 7
  Difference in Emotional Categorisation Task (ECAT): accuracy to classify positive and negative descriptor words
Change in reaction time in the Emotional Categorisation Task (ECAT) | Change between groups from baseline to day 7
  Differences in reaction time to classify positive and negative descriptor words
Change on Facial Dot Probe Task (FDOT) | Change between groups from baseline to day 7
  Differences in Vigilance scores derived from reaction time
Change on Emotional Recall Task (EREC) | Change between groups from baseline to day 7
  Differences in number of words correctly recalled (hits) and number of words incorrectly recalled (false alarms).
Change on Emotional Recognition Memory Task (EMEM) | Change between groups from baseline to day 7
  Difference in Emotional Recognition Memory Task (EMEM): accuracy and reaction time to correctly recognise positive and negative words (hits), and number of incorrectly recognised words (false alarms)
Change on brain inositol levels | Change between groups from baseline to day 7
  Difference in levels of inositol as determined by magnetic resonance spectroscopy (MRS)
Change on glutamate levels | Change between groups from baseline to day 7
  Difference in levels of glutamate as determined by MRS
Change on glutamine levels | Change between groups from baseline to day 7
  Difference in levels of glutamine as determined by MRS
Change on choline levels | Change between groups from baseline to day 7
  Difference in levels of choline as determined by MRS
Change in Montgomery-Åsberg Depression Rating scale (MADRS) | Change between groups from baseline to day 7
  Difference in the 10-item MADRS between groups. Total score 0-60.
Change in the Quick Inventory of Depressive Symptomatology-Self report (QIDS-SR) | Change between groups from baseline to day 7
  Difference in 16 item self-rated QIDS-SR between groups. Total score 0-42.
Change in Generalised Anxiety Disorder Assessment -7 (GAD-7) | Change between groups from baseline to day 7
  Difference in the 7 item self-rated GAD-7 between groups. Total score 0-21

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cowen, MBBS, MD, Principal Investigator — Dept. Psychiatry, University of Oxford
Locations (1):
- Neurosciences Building, Dept. Psychiatry, Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharpley AL, Williams C, Holder AA, Godlewska BR, Singh N, Shanyinde M, MacDonald O, Cowen PJ. A phase 2a randomised, double-blind, placebo-controlled, parallel-group, add-on clinical trial of ebselen (SPI-1005) as a novel treatment for mania or hypomania. Psychopharmacology (Berl). 2020 Dec;237(12):3773-3782. doi: 10.1007/s00213-020-05654-1. Epub 2020 Sep 9. PMID 32909076
- [Background] Singh N, Sharpley AL, Emir UE, Masaki C, Herzallah MM, Gluck MA, Sharp T, Harmer CJ, Vasudevan SR, Cowen PJ, Churchill GC. Effect of the Putative Lithium Mimetic Ebselen on Brain Myo-Inositol, Sleep, and Emotional Processing in Humans. Neuropsychopharmacology. 2016 Jun;41(7):1768-78. doi: 10.1038/npp.2015.343. Epub 2015 Nov 23. PMID 26593266
- [Background] Masaki C, Sharpley AL, Cooper CM, Godlewska BR, Singh N, Vasudevan SR, Harmer CJ, Churchill GC, Sharp T, Rogers RD, Cowen PJ. Effects of the potential lithium-mimetic, ebselen, on impulsivity and emotional processing. Psychopharmacology (Berl). 2016 Jul;233(14):2655-61. doi: 10.1007/s00213-016-4319-5. Epub 2016 Jun 2. PMID 27256357
- [Background] Masaki C, Sharpley AL, Godlewska BR, Berrington A, Hashimoto T, Singh N, Vasudevan SR, Emir UE, Churchill GC, Cowen PJ. Effects of the potential lithium-mimetic, ebselen, on brain neurochemistry: a magnetic resonance spectroscopy study at 7 tesla. Psychopharmacology (Berl). 2016 Mar;233(6):1097-104. doi: 10.1007/s00213-015-4189-2. Epub 2016 Jan 12. PMID 26758281
- [Background] Kil J, Lobarinas E, Spankovich C, Griffiths SK, Antonelli PJ, Lynch ED, Le Prell CG. Safety and efficacy of ebselen for the prevention of noise-induced hearing loss: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2017 Sep 2;390(10098):969-979. doi: 10.1016/S0140-6736(17)31791-9. Epub 2017 Jul 14. PMID 28716314